CLINICAL TRIAL: NCT02460562
Title: The Caries Prevention Effect of Surface Pre-reacted Glass-ionomer Filler Incorporated in Denture Base Resins on Edentulous Elderly People
Brief Title: Caries Prevention Effect of S-PRG Filler Incorporated in Denture Base Resins on Edentulous Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kritirat Kiatsirirote (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor-Investigator, Kritirat Kiatsirirote, Dentistry, Thammasat University
Organization: Thammasat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 67-4326
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Dental Caries
Keywords: resin denture base
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PMMA resin (Active Comparator): A denture base will be made with PMMA resin as a standard material.
  Interventions: Device: PMMA resin
- PMMA resin & S-PRG filler (Experimental): A denture base will be made from PMMA resin & S-PRG filler for subject to wear.
  Interventions: Device: S-PRG filler; Device: PMMA resin

INTERVENTIONS:
Device: S-PRG filler — Surface pre-reacted glass-ionomer (S-PRG) filler is a new type of biological material. This new material is being used in the formulation of dental product as filling materials. It has an anti-plaque effect which will release ions to alter the pH of the surrounding environment when it comes into contact with water or acidic solutions. These ions will exert their effect on caries prevention.
  The amount of S-PRG filler that is put in the standard resin denture base is 20% by weight. They are incorporated into the resin denture base and maintain the mechanical properties as required by ISO 1567.
  Other Names: Surface pre-reacted glass-ionomer filler
  Arms: PMMA resin & S-PRG filler
Device: PMMA resin — Polymethyl methacrylate (PMMA) resins have been used for the fabrication of resin denture base for 50 years. The advantages of PMMA resin that most notably is the ease of fabrication with very simple equipment but a limitation is the fragility because of its physical properties that include low flexural strength and surface hardness.
  Other Names: Polymethymethacrylate resin; resin denture base

SUMMARY:
The purpose of this study is to determine whether a novel material of S-PRG fillers containing in a daily-used resin denture base and their capability of fluoride release and recharge to elevate the salivary fluoride level and prevent dental caries in Thai middle-aged patients between 35-60 years of age who wear the resin denture.

DETAILED DESCRIPTION:
The study design is a 1.5-year, double blind randomized clinical trial, with 150 volunteers between 35-60 years of age wearing palatal removable partial denture containing with/without S-PRG fillers. This study will be performed in 3 local government hospitals located around Bangkok metropolitan, Ministry of Public Health, Thailand. The subjects will be assigned to the control group; resin denture base containing without S-PRG fillers and the experimental group; resin denture base containing 20% by weight of S-PRG fillers. Two parameters we can measure are; (1) Salivary fluoride level, accessed at different time point; on day 1, 14, 15 and at 3, 12 months after wearing the denture, and (2) Caries incidence using ICDAS-II, taken at 18 months.

Regarding an agreement with the participating dentists and dental assistants in the hospitals, patients in the waiting list of removable partial denture are screened according to our eligible criteria. If they meet eligibility criteria, a complete description is follow:

"If you agree to participate in the study, at today's visit we will ask you some questions about your medical and dental health such as what medication that you are presently taking, and whether you use fluoride supplement except for toothpaste. You do not have to answer every question. The dentist will do a brief examination of your mouth looking to see if you have any decay. You will not be able to participate in this study if you have obvious untreated tooth decay.

Following completion of the questionnaire and examination, we will do a simple test on your saliva. We will collect stimulated saliva by having you to chew a piece of wax for 5 minutes. You will spit all the saliva formed during those 5 minutes into a cup. We will measure the volume of the saliva produced. You will have to have a normal flow rate to participate.

Collecting this information, doing the saliva test, and completing the dental examination will take about 30 minutes of today's appointment. You may refuse to participate in any of the saliva test or answer any question or item in the questionnaire. If that is the case, you will not qualify for the study. If you do qualify and agree to take part, the dentist will take a mold of your mouth to make an upper resin denture to replace your missing teeth for you to wear. This is a routine dental procedure. Some subjects may gag while the mold is being taken for the denture. The dentist has methods to help you control the gagging reflex.

Depending on which group you are assigned, your resin denture will be made from standard material or the standard material containing some new type of biological material. This new material we are testing is being used in the formulation of dental product as filling materials.

At the next appointment, approximately two week later, you will come in to have the denture fitted for you. Slight discomfort may occur at the gum margin where the denture can pinch. The plate will be adjusted to relieve any pinching. On rare occasions, allergy to the resin denture base may occur. We will stop your participation in the study if you have an allergy to the resin denture.

We will give you the resin denture and need you to wear it all day excluding when you sleep at night. You must take it out to brush your teeth. You may clean the denture with water and the same toothbrush that you use to brush your teeth before keeping the denture in the denture storage box. We do not want you to use anything else on the denture except material we supply. You will receive a box for keeping your denture, toothbrush and toothpaste to brush your teeth at home.

At the first 14 days once you receive the denture, we do want you to soak your denture in a denture storage box containing tap water every night when you sleep. After that we will supply you a tube of fluoride gel for storing the denture instead of tap water. We will ask you to apply the gel (approximately 1 cm of length) to the denture and spread out totally on both side of the denture before keeping in the denture box during sleeping every night for 1.5 years.

After wearing the denture, you will be asked to return to the clinic for check-up and recall. We will collect your saliva while wearing the denture periodically for a total of six times within one year according to our schedule for the analysis of the fluoride level.

At 1.5 years, you will be asked to return to the clinic and the dentist will do a dental examination for follow-up. That will conclude your participation in the study.

We will assess the salivary fluoride at different time point during 1 year. The fluoride level of saliva will show us the capability of the new material on the fluoride release and recharge. The follow up period will be extended for 6 more months. The caries information collected at 1.5 years will show us the incidence of new caries. All procedures will be done at the dental clinic of the hospital. The subjects will be identified by a number assigned only. The principle investigator and the project coordinator will have to access to the code which will remain locked at all time. The saliva collected from the subjects will be discarded immediately after complete analysis.

The sample size assessment is considered based on the long term outcome, caries incidence, and the short term outcome, salivary fluoride concentration, of the study. The optimal sample size to address both outcomes in the study and allow for a 20% drop out rate would be 75 subjects per group (150 total) to provide sufficient statistical power to detect the difference in mean caries incidence between the control and the intervention group.

Collected data will be entered into a computer database and analyzed with STATA software version 12 for Windows. The statistical significance level will be set at α = 0.05.

The analysis plan for salivary fluoride level at each phase of follow up is based on two-sample t test and linear regression adjusting for confounders (age, number of remaining teeth).

Data analysis for caries incidence will be recorded per surface using ICDAS-II severity scores at 1.5 years. The caries outcome is defined as score 1 to 6 and 1 to 2 for root caries. Two-sample t test or linear regression with adjusting for age will be performed to assess the different between the control and the intervention group in the mean number of new surface caries (dmfs) ± standard deviations at 1.5 years follow-up examination.

ELIGIBILITY:
Inclusion Criteria:

* Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions
* General Health: Good general health with no clinically significant and/or relevant abnormalities of medical history or oral examination that could interfere with subject safety during the study period
* Salivary Flow: Have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate > 0.15 ml/minute; gum base stimulated saliva flow rate ≥ 1 ml/minute)
* Oral condition: a) At least 6 teeth remaining natural upper teeth in good condition, including at least 2 posterior teeth. b) Adequate remaining natural or artificial lower teeth for proper function. c) Do not use fluoride supplement excluding toothpaste. and d) Present of caries risk or filling at least 1 surface.

Exclusion Criteria:

* Exhibited signs of xerostomia
* Serious oral pathology (e.g. extensive dental caries, periodontal disease)
* Pregnant or lactating women
* Frequent mouthwash or fluoride supplement use
* Unable to have basic self-care ability (including oral hygiene practice)
* History of allergies, metabolic diseases such as diabetes, or other medical conditions that could interfere with the study.
* Be caries free in oral cavity

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08-30 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A DeRouen, PhD, Study Director — Forgaty International Center,NIH
Locations (3):
- Thailand (3):
  - Health Promotion Center 1, Bang Khen, Bangkok
  - Thammasat Hospital, Khlong Luang, Changwat Pathum Thani
  - Krathumbaen Hospital, Samut Sakhon, Samutsakorn

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kamijo K, Mukai Y, Tominaga T, Iwaya I, Fujino F, Hirata Y, Teranaka T. Fluoride release and recharge characteristics of denture base resins containing surface pre-reacted glass-ionomer filler. Dent Mater J. 2009 Mar;28(2):227-33. doi: 10.4012/dmj.28.227. PMID 19496404
- [Background] Mukai Y, Kamijo K, Fujino F, Hirata Y, Teranaka T, ten Cate JM. Effect of denture base-resin with prereacted glass-ionomer filler on dentin demineralization. Eur J Oral Sci. 2009 Dec;117(6):750-4. doi: 10.1111/j.1600-0722.2009.00678.x. PMID 20121940
- [Background] Ma S, Imazato S, Chen JH, Mayanagi G, Takahashi N, Ishimoto T, Nakano T. Effects of a coating resin containing S-PRG filler to prevent demineralization of root surfaces. Dent Mater J. 2012;31(6):909-15. doi: 10.4012/dmj.2012-061. PMID 23207194
- [Derived] Kiatsirirote K, Sitthisettapong T, Phantumvanit P, Chan DCN. Fluoride-Releasing Effect of a Modified Resin Denture Containing S-PRG Fillers on Salivary Fluoride Retention: A Randomized Clinical Study. Caries Res. 2019;53(2):137-144. doi: 10.1159/000490627. Epub 2018 Jul 27. PMID 30056451
- See also: Ion releasing by S-PRG filler — http://www.shofu.com/en/restoratives/187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of subjects was carried out through hospital media from three government hospitals; Krathum Baen Hospital, Samut Sakhon Province, Health Promotion Center Region 1, Bangkok and Thammasat University Hospital, Pathum Thani Province. Subjects who were interested in the study could register directly at the dental clinic.
Pre-assignment Details: Subjects who registered for a screening appointment at the dental clinic were asked to complete a questionnaire and underwent an oral screening and a simple test of salivary flow rate at the screening visit. The subjects who met eligibility criteria were asked whether or not they would agree to participate in the study.
Groups:
- PMMA Resin: A denture base was made with PMMA resin as a standard material.
  PMMA resin: Polymethyl methacrylate (PMMA) resins have been used for the fabrication of resin denture base for 50 years. The advantages of PMMA resin that most notably is the ease of fabrication with very simple equipment but a limitation is the fragility because of its physical properties that include low flexural strength and surface hardness.
- PMMA Resin & S-PRG Filler: A denture base was made from PMMA resin containing S-PRG fillers for subject to wear.
  Surface pre-reacted glass-ionomer (S-PRG) filler is a new type of biological material. This new material is being used in the formulation of dental product as filling materials. It has an anti-plaque effect which will release ions to alter the pH of the surrounding environment when it comes into contact with water or acidic solutions. These ions will exert their effect on caries prevention.
  The amount of S-PRG filler that is put in the standard resin denture base is 20% by weight. They are incorporated into the resin denture base and maintain the mechanical properties as required by ISO 1567.
  PMMA resin: Polymethyl methacrylate (PMMA) resins have been used for the fabrication of resin denture base for 50 years. The advantages of PMMA resin that most notably is the ease of fabrication with very simple equipment but a limitation is the fragility because of its physical properties that inc
Period: Overall Study
Arm/Group | PMMA Resin | PMMA Resin & S-PRG Filler
Started | 74 | 76
Completed | 59 | 60
Not Completed | 15 | 16
Not completed — Lost to Follow-up | 15 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PMMA Resin | PMMA Resin & S-PRG Filler | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 76 | 150
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.31 (10.81) | 47.66 (10.58) | 47.98 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 60 | 119
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  Thailand | 74 | 76 | 150

OUTCOME MEASURES:

1. Primary Outcome: Saliva Fluoride Concentration (Part Per Million,Ppm)
Description: Whole mixed saliva was collected by passive drooling into individual plastic vials to a volume of 2 ml while wearing the denture to determine the capacity for fluoride release and recharge from the denture. Saliva fluoride concentrations (ppm) were assessed at multiple time points (baseline, days 1, 14, 15, and 3 months and 1.5 years) to compare with baseline concentration under the conditions that the participants wear the resin denture at least 1 hour and refrain from tooth brushing at least 2 hours before saliva sampling. The salivary fluoride content (ppm) of each solution was determined using a fluoride ion electrode (item number 27502-19, Cole-Palmer, USA) connected to a 710 A plus fluoride ion meter (item number 067952, Thermo Orion, USA).
Time Frame: on days 1, 14, 15, and 3 months and 1.5 years of wearing the denture
Population: A total of 150 Thai adults aged 35-60 years, were initially enrolled in this study. At a baseline visit, 31 males (20.7%) and 119 females (79.3%) with a mean age of 48.9 ± 10.6 years fulfilled the study inclusion criteria and participated in this study. Approximately eighty percent (119/150) of the study adults were followed over 1.5 years.
Measure: Mean (Standard Deviation); unit: part per million,ppm
Groups:
- PMMA Resin & S-PRG Filler: A denture base was made from PMMA resin containing S-PRG fillers.
  Surface pre-reacted glass-ionomer (S-PRG) filler is a new type of biological material. This new material is being used in the formulation of dental product as filling materials. It has an anti-plaque effect which will release ions including fluoride to alter the pH of the surrounding environment when it comes into contact with water or acidic solutions. These ions will exert their effect on caries prevention.
  The amount of S-PRG filler that is put in the standard resin denture base is 20% by weight. They are incorporated into the resin denture base and maintain the mechanical properties as required by ISO 1567.
Arm/Group | PMMA Resin | PMMA Resin & S-PRG Filler
Number analyzed (Participants) | 74 | 76
part per million,ppm
  Baseline | 0.05 (0.04) | 0.05 (0.05)
  Day 1 | 0.09 (0.07) | 0.22 (0.12)
  Day 14 | 0.06 (0.06) | 0.06 (0.05)
  Day 15 | 0.11 (0.11) | 0.23 (0.13)
  3 months | 0.12 (0.12) | 0.26 (0.15)
  1.5 Years | 0.08 (0.12) | 0.32 (0.2)
Statistical Analysis 1: Comparison: PMMA Resin vs PMMA Resin & S-PRG Filler; Mean saliva fluoride concentration (part per million) collected at different time points was compared in order to assess the change in capacity for fluoride release and recharge from the resin denture base and to assess differences between the control and the intervention group; Test type: Superiority; p < 0.05, ANOVA — Mean salivary fluoride concentrations (part per million) between groups were assessed at different time points using repeated measures analysis of variance. Saliva fluoride concentration from each groups were compared with baseline using a t-test

2. Secondary Outcome: Assessment of Enamel Caries
Description: Caries record per surface using ICDAS coding system were determined at baseline and at 1.5 years of follow-up
Time Frame: Baseline and 1.5 years of follow up
Population: The transition (∆Q) of surface number, n (%) of developed new caries from baseline to 1.5 years of follow up was determined as progression or arrested rate.
Measure: Count of Units; unit: Caries examined (number of surface)
Units Other Than Participants: Caries examined (number of surface)
Arm/Group | PMMA Resin | PMMA Resin & S-PRG Filler
Number analyzed (Participants) | 74 | 76
Number analyzed (Caries examined (number of surface)) | 3523 | 3479
Caries examined (number of surface)
  Arrest | 3353 | 3402
  Progress | 170 | 77
Statistical Analysis 1: Comparison: PMMA Resin vs PMMA Resin & S-PRG Filler; Caries assessments were performed to examine the difference in mean number of surface caries (DMFS) ± standard deviation between the control and the intervention groups at baseline and at 1.5 years.The transition (∆Q) of developed new caries surfaces (ICDAS score 1-3) from baseline to 1.5 years of follow-up for the two groups was analyzed with respect to arrest or progress rates. Numbers of new caries surfaces were compared by independent t-test, Pearson chi-square and correlation coefficient; Test type: Superiority; p < 0.05, Chi-squared; Odds Ratio (OR) = 0.45

ADVERSE EVENTS:
Time Frame: The study was followed for 1.5 years. This period of time collected for adverse event data.
Description: Adverse event were assessed and monitored during the study. However, no adverse event was found.
Arm/Group | PMMA Resin | PMMA Resin & S-PRG Filler
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/76
Other Adverse Events (participants affected / at risk) | 0/74 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No